CLINICAL TRIAL: NCT01136083
Title: Effect of Exercise Training on Angiogenesis and Cachexia in Lung Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201003064R
Record Dates: First submitted 2010-05-10; First posted 2010-06-03 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2011-11

CONDITIONS: Non-small-cell Lung Cancer
Keywords: Tumor; Angiogenesis; Exercise training; VEGF; Myostatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Exercise; Patient Education as Topic

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise training (Experimental): Subjects in exercise group will undergo individualized high aerobic interval training on treadmill for 30 minutes under the supervision of an experienced physical therapist 3 times a week and home exercise twice a week with accelerometer.
  Interventions: Behavioral: Exercise training
- Control group (Active Comparator): Subjects in control group will not undergo individualized high aerobic interval training on treadmill. They will receive usual care as normally does in hospital.
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Exercise training — Subjects in exercise group will undergo individualized high aerobic interval training on treadmill for 30 minutes under the supervision of an experienced physical therapist 3 times a week and home exercise twice a week with accelerometer.
  Other Names: High intensity interval aerobic training
  Arms: Exercise training
Other: Usual care — Subjects in control group will not undergo individualized high aerobic interval training on treadmill. They will receive usual care as normally does in hospital.
  Other Names: Non-exercise or patient education
  Arms: Control group

SUMMARY:
Cancer is one of the leading health issues in this country and worldwide. Angiogenesis is an essential process for tumoral growth and metastasis. This process is dependent on the balance between angiogenic factors and antiangiogenic factors. Muscle wasting has been associated with myostatin overexpression in cancer. Exercise training can depress tumor growth and suppress myostatin expression, and enhance skeletal muscle angiogenesis in healthy people and some animal studies. The purpose of this study is mainly to investigate the effects of exercise training on

1. circulating VEGF-A
2. muscle growth and function
3. Myostatin

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75 years
* Advanced NSCLC
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Targeted therapy for at least 8 weeks
* Stable condition

Exclusion Criteria:

* Severe metastasis, cardiopulmonary or musculoskeletal conditions may affect participation in exercise
* Do not understand the verbal or written instructions

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Exercise capacity | 8 weeks after the start of the intervention
  Maximal oxygen consumption with Vmax229 Vastus lateral muscle oxygenation with NIRS

SECONDARY OUTCOMES:
Imaging of muscle | 8 weeks and 16 weeks after the start of the intervention
  Measured by MRS
Analysis of venous blood sample | 8 weeks andd 16 weeks after the start of the intervention
  Analysis of circulating VEGF-A and myostatin
Quality of life | baseline, 8 weeks, 16 weeks
  Measured by questionnaire
Exercise capacity | 16 weeks after the start of the intervention
  Maximal oxygen consumption with Vmax229 Vastus lateral muscle oxygenation with NIRS
Muscle function | 8 weeks and 16 weeks after the start of the intervention
  Isokinetic muscle strength and endurance with Biodex
Physical activity | 8 weeks andd 16 weeks after the start of the intervention
  Measured with 7-day recall questionnaire
Dietary intake | 8 weeks andd 16 weeks after the start of the intervention
  Measured with 24-hour recall questionnaire
Body composition | 8 weeks andd 16 weeks after the start of the intervention
  Body mass index calculated with body weight and height
  % body fat abd free-fat mass with BIA

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Tai Wu, Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan